CLINICAL TRIAL: NCT02521077
Title: Prospective Double Blind Study of the Effect of Intravenous High Dose Ascorbic Acid in Women Receiving Adjuvant or Neo-Adjuvant Chemotherapy for Early Stage Breast Cancer
Brief Title: Intravenous Ascorbic Acid in Women Receiving Adjuvant or Neo-Adjuvant Chemotherapy for Early Stage Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer unwilling to provide information needed for IND application.
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Citrin, MD, Medical Oncologist, Midwestern Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MZ2015010
Record Dates: First submitted 2015-07-27; First posted 2015-08-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Fatigue
Keywords: Ascorbic Acid; Breast Neoplasms; Fatigue
MeSH Terms: conditions — Fatigue; Breast Neoplasms | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Odd Cycle Intravenous Ascorbic Acid (Experimental): Women randomized to this study arm will receive intravenous ascorbic acid (50g in 500 ml sterile water) prior to their odd-numbered chemotherapy cycles. During the even-numbered chemotherapy cycles, these subjects will receive intravenous normal saline (0.9%).
  Interventions: Drug: Ascorbic Acid; Other: Normal Saline
- Even Cycle Intravenous Ascorbic Acid (Experimental): Women randomized to this study arm will receive intravenous ascorbic acid (50g in 500 ml sterile water) prior to their even-numbered chemotherapy cycles. During the odd-numbered chemotherapy cycles, these subjects will receive intravenous normal saline (0.9%).
  Interventions: Drug: Ascorbic Acid; Other: Normal Saline

INTERVENTIONS:
Drug: Ascorbic Acid — 500 g ascorbic acid dissolved in 500 ml sterile water.
  Other Names: Vitamin C
Other: Normal Saline — Saline 0.9%

SUMMARY:
This is a parallel-track, randomized study will observe whether intravenous ascorbic acid reduces the reported fatigue in women receiving adjuvant or neo-adjuvant chemotherapy for early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
* Diagnosed early stage breast cancer and scheduled to receive either adjuvant or neo-adjuvant chemotherapy;
* Willing to receive either intravenous ascorbic acid or normal saline;
* Willing to use an acceptable contraceptive method for the duration of the study and for 30 days following the last dose of study drug;
* Negative urine or serum pregnancy test within 2 weeks prior to receipt of study drug;
* Willing to complete all evaluation tools;
* Able to give informed consent to participate in the study; and
* Agree to avoid any additional supplemental ascorbic acid throughout the study.

Exclusion Criteria:

* Diagnosed Glucose-6-phosphate dehydrogenase deficiency;
* Renal insufficiency (Blood Urea Nitrogen >30 mg/dL, or Creatinine >1.5 mg/dL);
* Unwillingness or mental incapacity to complete self-reported questionnaires;
* Active smoker; and
* Male sex

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue by self reported fatigue inventory questionnaire | Day 8 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire Fatigue Symptom Inventory (FSI)

SECONDARY OUTCOMES:
Fatigue ( EORTC QLQ-FA13) | Day 1 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire EORTC QLQ-FA13
Fatigue ( EORTC QLQ-FA13) | Day 8 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire EORTC QLQ-FA13
Fatigue ( EORTC QLQ-FA13) | Day 15 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire EORTC QLQ-FA13
Fatigue by self reported fatigue inventory questionnaire | Day 1 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire Fatigue Symptom Inventory (FSI)
Fatigue by self reported fatigue inventory questionnaire | Day 15 of each 4-week treatment cycle.
  Patients will complete the validated questionnaire Fatigue Symptom Inventory (FSI)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Citrin, MD, PhD, Principal Investigator — Midwestern Regional Medical Center